CLINICAL TRIAL: NCT03311633
Title: Distal Radius Fracture: Comparison Between Three and Six Weeks of Percutaneous Fixation
Brief Title: Complications in Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos A Acosta-Olivo (Other)
Responsible Party: Sponsor-Investigator, Carlos A Acosta-Olivo, Principal Investigator, Universidad Autonoma de Nuevo Leon
Organization: Universidad Autonoma de Nuevo Leon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR17-00011
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Radius Fracture Distal
Keywords: Radius Fracture Distal; Radius Fracture Distal Therapy; Fracture fixation; Closed Fracture Reduction
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Three week percutaneous pinning group versus Six week percutaneous pinning group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 week percutaneous pinning group (Experimental): Percutaneous pinning time will be for three weeks and short cast immobilization for six weeks.
  Interventions: Procedure: Percutaneous pinning time
- 6 week percutaneous pinning group (Active Comparator): Percutaneous pinning time will be for six weeks and also short cast immobilization.
  Interventions: Procedure: Percutaneous pinning time

INTERVENTIONS:
Procedure: Percutaneous pinning time — Percutaneous pinning time will be compared in two groups: 3 versus 6 weeks.

SUMMARY:
BACKGROUND. Distal radius fractures (FRD) are up to 17% of all diagnosed fractures and are the most commonly treated fractures in adult orthopedic patients. The management could be either conservative or surgical, depending on AO bone fracture classification. The principles of good treatment involves an anatomical reduction with a proper immobilization that keep the reduction.

OBJECTIVE. Determine if percutaneous pinning for six weeks versus three has major complications in distal radius fractures.

DETAILED DESCRIPTION:
Distal radius fractures (DRF) are up to 20% of all diagnosed fractures and are the most commonly treated fractures in adult orthopedic patients. DRF occur in distal third of the radius bone, located less than 2.5 cm from the radiocarpal joint. In general, it is the result of a fall on the hand in extension. A bimodal distribution is observed with a peak incidence predominantly in young adult patients and another peak in elderly women. In the younger population these fractures are usually the result of high-impact injuries such as vehicular accidents or high-altitude falls. This diagnosis in elderly most commonly occurs by falls from their own height and other low-energy trauma.

The management could be either conservative or surgical, depending on AO bone fracture classification. Regarding treatment, there is still much controversy as to what procedure would be ideal in each case. When selecting the therapeutic method, the patient's age, work, functional status and daily activities should be considered. Therapeutic alternatives differ considerably around the world and no technique has proven to be superior to all others, and there is no particular method that yields acceptable results in all types of DRF. The principles of good treatment involves an anatomical reduction with a proper immobilization that keep the reduction.

If segmental or unstable fractures are not treated properly, serious complications can occur. The rate of complications reported in the literature varies from 6 to 80% and these may be a consequence of the fracture or its treatment. There are many vital structures of soft tissue in close proximity to the bony anatomy around the wrist and the complications associated with these soft tissues may be more problematic than the fracture. Some surgical complications are loss of mobility, delayed consolidation, pseudoarthrosis, nerve compression, painful syndromes, complications of fixation material, osteomyelitis, vicious consolidation, tendon rupture, tenosynovitis, pathological scarring, radio-cubital synostosis, Dupuytren's contracture, arthritis and ligament injury. However, cutaneous complications such as ulcers or granulomas may occur at the site of nails, although not usually serious complications may prevent early rehabilitation of the patient and extend recovery times for incorporation into their daily activities.

Statistical analysis. The results will be reported in contingency tables, frequencies, percentages, measures of central tendency and dispersion. Qualitative variables will be analyzed with the chi-square statistic and quantitative variables with t-test for independent samples with a significance level of 95% with their respective confidence intervals, or with non-parametric statistics if necessary. Using a mean difference formula with a standard deviation of 5 and an expected magnitude of the differences of at least 4 points on the PRWE scale, with a confidence interval of 95%, a power β of 80%, with a statistically significant p = ˂0.05, adding 20% of error. A sample of 30 participants was obtained per group. For evaluation of pain (Visual Analogue Scale) and functional evaluation (Patient Rated Wrist Evaluation), the Student's T test and one-way ANOVA with Tuckey's post-hoc test will be performed for multiple comparisons in order to identify differences between groups. Statistical analysis will be performed with IBM SPSS version 20 (SPSS, Inc., Armon, NY).

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 ages
* any gender
* distal radius fracture type A or B of AO classification managed with closed reduction and percutaneous pinning
* and Informed Consent signature

Exclusion Criteria:

* associated ipsilateral fractures in the upper extremity
* fractures attended and fixed at another institution
* support external fixation
* previous skin conditions (infection, ulcers)
* limitation of wrist mobility prior to injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 14 week
  It´s a numeric scale, when 0 value is equal to no pain; and 10 is equal to a maximum pain

SECONDARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | 14 weeks
  It´s a 15- item questionnaire designed to measure wrist pain and disability in activities of daily living. developed in 1998 for clinical assessment and is used for specific wrist problems. It is one of the reliable upper extremity outcome instrument
Wrist mobility | 14 weeks
  Mobility in flexion, extension, pronation, supination, cubital and radial deviation using a goniometer.
Grip strength | 14 weeks
  Using a hydraulic dynamometer with the patient's elbow in 90 grades of flexion and forearm in neutral rotation.
Skin condition | 6 weeks
  Evaluation of skin condition and integrity, when normal is equal to 0, ulcer=1 and granuloma=2

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided

REFERENCES:
- [Result] Tahririan MA, Javdan M, Motififard M. Results of pronator quadratus repair in distal radius fractures to prevent tendon ruptures. Indian J Orthop. 2014 Jul;48(4):399-403. doi: 10.4103/0019-5413.136275. PMID 25143645
- [Result] Niver GE, Ilyas AM. Carpal tunnel syndrome after distal radius fracture. Orthop Clin North Am. 2012 Oct;43(4):521-7. doi: 10.1016/j.ocl.2012.07.021. Epub 2012 Sep 4. PMID 23026468
- [Result] Dhainaut A, Daibes K, Odinsson A, Hoff M, Syversen U, Haugeberg G. Exploring the relationship between bone density and severity of distal radius fragility fracture in women. J Orthop Surg Res. 2014 Jul 17;9:57. doi: 10.1186/s13018-014-0057-8. PMID 25030810
- [Result] Henn CM, Wolfe SW. Distal radius fractures in athletes: approaches and treatment considerations. Sports Med Arthrosc Rev. 2014 Mar;22(1):29-38. doi: 10.1097/JSA.0000000000000003. PMID 24651288
- [Result] Turner RG, Faber KJ, Athwal GS. Complications of distal radius fractures. Orthop Clin North Am. 2007 Apr;38(2):217-28, vi. doi: 10.1016/j.ocl.2007.02.002. PMID 17560404
- [Result] Davis DI, Baratz M. Soft tissue complications of distal radius fractures. Hand Clin. 2010 May;26(2):229-35. doi: 10.1016/j.hcl.2009.11.002. PMID 20494749